CLINICAL TRIAL: NCT01212640
Title: GROUP FOR TRALI STUDY. SEMICYUC.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Hospitales Universitarios Virgen del Rocío (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Germans Trias i Pujol Hospital (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Dr. Negrin University Hospital (Other); Hospital Universitari Son Dureta (Other); Hospital Miguel Servet (Other)
Responsible Party: CARMEN MARIA FERRANDIZ MILLON, FISEVI
Other Study IDs: TRALI STUDY. SEMICYUC
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2010-09

CONDITIONS: Acute Lung Injury
Keywords: Transfusion, distress
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
OBJETIVES:

1. To research the worsening of respiratory status risk factors after transfusion in spanish critical care units.
2. To determine the incidence of transfusion-related acute lung injury (TRALI) in critically ill patients.
3. To research the morbi-mortality of TRALI.

DETAILED DESCRIPTION:
Actually there are no published European data on the incidence of acute lung injury by transfusion (TRALI) in critically ill patients, in Europe, estimates of TRALI incidence are limited to passive reports of national blood banks. This multicenter study of Spanish ICUs will investigate the incidence and TRALI predisposing factors (associated with the patient, the transfused blood product and the presence or absence of mechanical ventilation).

Design:

Prospective multicenter observational study.

Patients:

All patients transfused in eleven spanish intensive care units (UCI) from October 1, until November 30, 2010. Patients with less of 18 years old, or transfused six hours before be included in this study or seriousness patients with a length of stay <24 hrs will be excluded.

Variables:

* Patient data collection: Demografic data (age, gender), Clinical data (comorbid conditions), Admission diagnostic , Complications during the stay and severity of illness scores: Acute Physiology and Chronic Health Evaluation (APACHE II) score, Sequential Organ Failure Assessment (SOFA) score, Euroscore.
* Transfusion factors: Type of blood product, time of infusion and volumen transfused, storage age and donor sex.
* Respiratory factors: Main ventilation and oxigenation parameters and type of respiratory support before and after transfusion.

For each transfusion episode was completed two data tables (see last page of the booklet of data collection):

* Before the transfusion (baseline) are listed the values of the patient's respiratory function, the analytical value that is transfused (Hb, INR, APTT, PT, platelets) and the number of the bag that is transfused (to apply blood bank storage time and sex of the donor).
* After the transfusion are recorded the volume and time infusion and 6 hours after transfusion are collected again the parameters of the patient's respiratory function and radiographic changes.

According to official criteria shall be noted if the patient has exhibited a classic TRALI, possible TRALI, or a worsening of their respiratory function after transfusion.

ELIGIBILITY:
Inclusion Criteria:

* All patients transfused in eleven spanish intensive care units (UCI) from October 1, until November 30, 2010.

Exclusion Criteria:

* Patients with less of 18 years old, or transfused six hours before be included in this study or seriousness patients with a length of stay <24 hrs will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients transfused in eleven spanish intensive care units (UCI) from October 1, until November 30, 2010. Patients with less of 18 years old, or transfused six hours before be included in this study or seriousness patients with a length of stay <24 hrs will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Worsening of respiratory status | October-November
  To research the worsening of respiratory status risk factors after transfusion in spanish critical care units.

SECONDARY OUTCOMES:
Incidence and morbi-mortality of TRALI | October-November
  Determine the incidence and morbi-mortality of transfusion-related acute lung injury (TRALI) in critically ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: CARMEN MARIA FERRANDIZ, MD, Principal Investigator
Locations (2):
- Spain (2):
  - Hospital Virgen Del Rocio, Seville, Sevilla
  - Hospital Virgen Del Rocio, Seville, Seville

REFERENCES:
- [Background] Silliman CC, Fung YL, Ball JB, Khan SY. Transfusion-related acute lung injury (TRALI): current concepts and misconceptions. Blood Rev. 2009 Nov;23(6):245-55. doi: 10.1016/j.blre.2009.07.005. Epub 2009 Aug 20. PMID 19699017
- [Background] Toy P, Popovsky MA, Abraham E, Ambruso DR, Holness LG, Kopko PM, McFarland JG, Nathens AB, Silliman CC, Stroncek D; National Heart, Lung and Blood Institute Working Group on TRALI. Transfusion-related acute lung injury: definition and review. Crit Care Med. 2005 Apr;33(4):721-6. doi: 10.1097/01.ccm.0000159849.94750.51. PMID 15818095
- [Background] Goldman M, Webert KE, Arnold DM, Freedman J, Hannon J, Blajchman MA; TRALI Consensus Panel. Proceedings of a consensus conference: towards an understanding of TRALI. Transfus Med Rev. 2005 Jan;19(1):2-31. doi: 10.1016/j.tmrv.2004.10.001. PMID 15830325
- [Background] Gajic O, Rana R, Winters JL, Yilmaz M, Mendez JL, Rickman OB, O'Byrne MM, Evenson LK, Malinchoc M, DeGoey SR, Afessa B, Hubmayr RD, Moore SB. Transfusion-related acute lung injury in the critically ill: prospective nested case-control study. Am J Respir Crit Care Med. 2007 Nov 1;176(9):886-91. doi: 10.1164/rccm.200702-271OC. Epub 2007 Jul 12. PMID 17626910
- [Background] Gong MN, Thompson BT, Williams P, Pothier L, Boyce PD, Christiani DC. Clinical predictors of and mortality in acute respiratory distress syndrome: potential role of red cell transfusion. Crit Care Med. 2005 Jun;33(6):1191-8. doi: 10.1097/01.ccm.0000165566.82925.14. PMID 15942330
- [Background] Eder AF, Benjamin RJ. TRALI risk reduction: donor and component management strategies. J Clin Apher. 2009;24(3):122-9. doi: 10.1002/jca.20198. PMID 19365816
- [Background] Yilmaz M, Keegan MT, Iscimen R, Afessa B, Buck CF, Hubmayr RD, Gajic O. Toward the prevention of acute lung injury: protocol-guided limitation of large tidal volume ventilation and inappropriate transfusion. Crit Care Med. 2007 Jul;35(7):1660-6; quiz 1667. doi: 10.1097/01.CCM.0000269037.66955.F0. PMID 17507824
- [Background] Benson AB, Moss M, Silliman CC. Transfusion-related acute lung injury (TRALI): a clinical review with emphasis on the critically ill. Br J Haematol. 2009 Nov;147(4):431-43. doi: 10.1111/j.1365-2141.2009.07840.x. Epub 2009 Aug 5. PMID 19663827
- [Background] Zilberberg MD, Carter C, Lefebvre P, Raut M, Vekeman F, Duh MS, Shorr AF. Red blood cell transfusions and the risk of acute respiratory distress syndrome among the critically ill: a cohort study. Crit Care. 2007;11(3):R63. doi: 10.1186/cc5934. PMID 17553147
- [Background] Chaiwat O, Lang JD, Vavilala MS, Wang J, MacKenzie EJ, Jurkovich GJ, Rivara FP. Early packed red blood cell transfusion and acute respiratory distress syndrome after trauma. Anesthesiology. 2009 Feb;110(2):351-60. doi: 10.1097/ALN.0b013e3181948a97. PMID 19164959
- [Background] Silverboard H, Aisiku I, Martin GS, Adams M, Rozycki G, Moss M. The role of acute blood transfusion in the development of acute respiratory distress syndrome in patients with severe trauma. J Trauma. 2005 Sep;59(3):717-23. PMID 16361918
- [Background] Vlaar AP, Binnekade JM, Prins D, van Stein D, Hofstra JJ, Schultz MJ, Juffermans NP. Risk factors and outcome of transfusion-related acute lung injury in the critically ill: a nested case-control study. Crit Care Med. 2010 Mar;38(3):771-8. doi: 10.1097/CCM.0b013e3181cc4d4b. PMID 20035217
- [Background] Williamson LM, Lowe S, Love EM, Cohen H, Soldan K, McClelland DB, Skacel P, Barbara JA. Serious hazards of transfusion (SHOT) initiative: analysis of the first two annual reports. BMJ. 1999 Jul 3;319(7201):16-9. doi: 10.1136/bmj.319.7201.16. PMID 10390452
- [Background] Wiersum-Osselton JC, Porcelijn L, van Stein D, Vlaar AP, Beckers EA, Schipperus MR. [Transfusion-related acute lung injury (TRALI) in the Netherlands in 2002-2005]. Ned Tijdschr Geneeskd. 2008 Aug 9;152(32):1784-8. Dutch. PMID 18754313
- [Background] Rebibo D, Hauser L, Slimani A, Herve P, Andreu G. The French Haemovigilance System: organization and results for 2003. Transfus Apher Sci. 2004 Oct;31(2):145-53. doi: 10.1016/j.transci.2004.07.010. PMID 15501418